CLINICAL TRIAL: NCT00046462
Title: Substituting Lantus®(Insulin Glargine[rDNAorigin]Inj) for a Thiazolidinedione vs. a 3rd Oral Agent as add-on Therapy in Patients Failing a Thiazolidinedione & Sulfonylurea or Metformin Combination
Brief Title: Determine Whether Glycemic Control is Different Between Lantus & a 3rd Oral Agent When Failure With Other Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_4022
Record Dates: First submitted 2002-09-30; First posted 2002-10-02 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Glargine; Injections; Metformin; Glyburide; 2,4-thiazolidinedione

INTERVENTIONS:
Drug: Lantus (insulin glargine [rDNA origin] injection)
Drug: Metformin
Drug: Glyburide
Drug: Thiazolidinedione

SUMMARY:
The purposes of the study is to determine whether blood sugar control is different between Lantus and a third oral anti-diabetic agent when added to patients who fail a thiazolidinedione and sulfonylurea or metformin combination.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 - 79 years of age
* With diagnosed type 2 diabetes for at least a year treated with stable doses of two oral antidiabetic drugs of which one is either Avandia or Actos for at least three months

Exclusion Criteria:

* Major cardiovascular events

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2001-11; Primary Completion 2004-11 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
To determine the difference in glycemic control as measured by HbA1C between substituting the TZD with insulin glargine and adding a third oral agent in patients who fail a TZD/sulfonylurea or TZD/metformin combination therapy | During the Study Conduct

SECONDARY OUTCOMES:
Occurrence of hypoglycemia | During the study conduct
Change in fasting plasma glucose | During the study conduct
Percentage of patients achieving HbA1C less than or equal to 7% | During the study conduct
Time to glycemic control | During the study conduct
Change in body weight | During the study conduct
Change in serum lipid profile | During the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Doug Green, Study Director — Sanofi
Locations (1):
- Aventis, Bridgewater, New Jersey, United States

REFERENCES:
- [Derived] Hollander P, Sugimoto D, Vlajnic A, Kilo C. Combination therapy with insulin glargine plus metformin but not insulin glargine plus sulfonylurea provides similar glycemic control to triple oral combination therapy in patients with type 2 diabetes uncontrolled with dual oral agent therapy. J Diabetes Complications. 2015 Nov-Dec;29(8):1266-71. doi: 10.1016/j.jdiacomp.2015.05.022. Epub 2015 Jun 5. PMID 26281972